CLINICAL TRIAL: NCT03020914
Title: Effects of Audiovisual Distraction Versus Standard Sedation on Desaturation and Airway Intervention in OSA-patients Undergoing Total Knee Arthroplasty Under Neuraxial Anesthesia
Brief Title: Effects of Audiovisual Distraction on Desaturation and Airway Intervention in OSA-patients
Acronym: AVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-0648
Record Dates: First submitted 2017-01-04; First posted 2017-01-13 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Audiovisual Distraction (Experimental): Patients get audiovisual distraction during surgery and in the recovery room using video goggles and headphones; patients can choose a movie from a preexisting library; with an initial dose of midazolam in preparation for the administration of the neuraxial anesthesia, additional sedation with midazolam in 1 mg increments if requested by the patient or deemed necessary by the anesthesia provider.
  Interventions: Device: Audiovisual Distraction
- Standard of care sedation (No Intervention): Standard of care sedation with with a initial dose of midazolam in preparation for the administration of the neuraxial anesthesia; propofol infusion titrated to effect.

INTERVENTIONS:
Device: Audiovisual Distraction — watching a movie using video glasses and headphones
  Other Names: Audiovisual Aids; Zeiss Cinemizer OLED Glasses; HappyMed Video Glasses
  Arms: Audiovisual Distraction

SUMMARY:
Patients will be randomly assigned to either one of two groups:

1. Standard of care sedation
2. Audiovisual distraction during surgery and in the recovery room using video goggles and headphones; patients can choose a movie from a preexisting library

Monitoring and anesthesia regimen will be standardized

DETAILED DESCRIPTION:
Before consent patients will be thoroughly informed about possible risks or benefits and about their possibilities to end the study at any time point or to ask for additional sedation if they feel uncomfortable or anxious. After they consent, they will be randomly assigned to either receive standard sedation (Group 1) or audiovisual distraction (Group 2). Each group will consist of 30 patients. The randomization schedule will be created by a member of the Healthcare Research Institute using SAS software, who is not otherwise involved in the trial.

1. Standard of care sedation with an initial dose of midazolam in preparation for the administration of the neuraxial anesthesia; propofol infusion titrated to effect.
2. Audiovisual distraction during surgery and in the recovery room using video goggles and headphones; patients can choose a movie from a preexisting library; with an initial dose of midazolam in preparation for the administration of the neuraxial anesthesia, additional sedation with midazolam in 1 mg increments if requested by the patient or deemed necessary by the anesthesia provider.

The intraoperative anesthesia regimen will be standardized:

* All patients will be monitored according to the American Society of Anesthesiologists standard, receive either a radial arterial line or non-invasive blood pressure measurement according to the preferences of the anesthesia provider and O2 via nasal cannula or face mask in the operation room and the recovery room.
* ondansetron,decadron and ketorolac may be administered as per clinical judgment of the attending anesthesiologist.
* Patients in both groups will receive neuraxial anesthesia. The attending anesthesiologist is free to add an ultrasound guided peripheral nerve block:

  * Neuraxial anesthesia (combined spinal-epidural, epidural or spinal) as preferred by the attending anesthesiologist. Decadron may be used as in addition to the local anesthetic if the anesthesia provider wishes to do so.
  * If a peripheral nerve block is performed the appropriate amount of bupivacaine will be administered under ultrasound-guidance as a single shot.
  * In case an epidural catheter was placed patients will receive a patient controlled epidural analgesia immediately after arrival at the recovery room for postoperative pain management.
* Opioids and other medications with sedative or respiratory depressant side effects that are not specifically mentioned above should be omitted (if possible without harm for the patient) Patients in the audiovisual distraction group will choose a movie, start watching it in the holding area and continue watching it in the operation room as well as the first 30 min in the recovery room. Audiovisual equipment will be removed for transfers or at patient request.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known OSA (preexisting diagnosis of obstructive sleep apnea (OSA) or patients with a STOP BANG Score of 5 or above) undergoing primary total knee arthroplasty under neuraxial anesthesia

Exclusion Criteria:

* Contraindications to neuraxial anesthesia or allergy to study medication
* Patients with audiovisual impairments prohibiting them from proper use of the study device:
* Patients who are blind
* Patients with hearing aids
* Age <18 years
* Patients with inability to communicate in English or understand the study requirements
* Patients with prior history of claustrophobia
* Patients with prior history of epilepsy or seizure disorder
* Patients undergoing a revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros G Memtsoudis, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Audiovisual Distraction | Standard of Care Sedation
Started | 10 | 9
Completed | 9 | 9
Not Completed | 1 | 0
Not completed — Surgery Cancelled | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Audiovisual Distraction | Standard of Care Sedation | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.04) | 69 (4.70) | 66 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Desaturations
Description: number of desaturation events (SpO2< 90% for ≥ 10 sec) measured during this time frame
Time Frame: start of anesthesia until 30 minutes after recovery room admission (ca. 3 hours)
Measure: Median (Inter-Quartile Range); unit: number of desaturation events
Arm/Group | Audiovisual Distraction | Standard of Care Sedation
Number analyzed (Participants) | 9 | 9
number of desaturation events | 0 [0 to 0] | 1 [0 to 1]

2. Secondary Outcome: Airway Interventions
Description: each airway intervention (defined as one of the following: jaw thrust, oropharyngeal airway, nasopharyngeal airway, mask ventilation, larynx mask or intubation) that is implemented during this time frame will be observed and documented by research staff, if it occurs.
Time Frame: start of anesthesia until 30 minutes after recovery room admission (ca. 3 hours)
Measure: Number; unit: airway interventions
Arm/Group | Audiovisual Distraction | Standard of Care Sedation
Number analyzed (Participants) | 9 | 9
airway interventions | 2 | 7

3. Secondary Outcome: Additional Sedation
Description: Patient request for additional sedation
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Audiovisual Distraction | Standard of Care Sedation
Number analyzed (Participants) | 9 | 9
Participants | 2 | 1

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction at recovery room discharge as measured by the Heidelberg perianesthetic questionnaire, which assesses patients' peri-anaesthetic satisfaction on a four-point Likert scale ranging from 0 (unimportant to me) to 3 (very important to me). Scores for each question are summed for a final score, with higher total score signifying higher satisfaction and lower total score signifying lower satisfaction. The score scale has a minimum value of 0 and a maximum value of 114 (based off 3 as the highest response score for 38 individual questions).
Time Frame: 10 minutes before recovery room discharge
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Audiovisual Distraction | Standard of Care Sedation
Number analyzed (Participants) | 9 | 9
score on a scale | 55 [49 to 56] | 54 [50 to 56]

5. Secondary Outcome: Alertness Levels
Description: Alertness levels measured using the Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/S), which rates alertness on a scale of 0-5, with higher ratings representing increased alertness (e.g. '5 - Responds readily to name spoken in normal tone'). Results reflect a median score of ratings collected at 4 time points.
Time Frame: 4 times: preoperative, intraoperative, at time of recovery room admission, 10 minutes before recovery room discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Audiovisual Distraction | Standard of Care Sedation
Number analyzed (Participants) | 9 | 9
score on a scale | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: All-cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: All-cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Audiovisual Distraction | Standard of Care Sedation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03020914/Prot_SAP_000.pdf